CLINICAL TRIAL: NCT07025785
Title: Molecular Residual Disease Assessment in a Representative Diverse Population of Patients With Early-stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Haystack Oncology, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC2412-DCT
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Lymph Node Metastasis
Keywords: circulating tumor DNA (ctDNA); minimal residual disease (MRD); African American
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1:Non African American (Experimental): 50 Non-African American participants with lymph node-positive (1-3 LNs) early breast cancer (all subtypes).
  Interventions: Diagnostic Test: Circulating tumor DNA
- 2: African American (Experimental): 50 African American participants with lymph node-positive (1-3 LNs) early breast cancer (all subtypes).
  Interventions: Diagnostic Test: Circulating tumor DNA

INTERVENTIONS:
Diagnostic Test: Circulating tumor DNA — Circulating tumor DNA (ctDNA) is a noninvasive prognostic biomarker for disease monitoring. ). Blood collection for ctDNA testing will be performed at the time of enrollment (prior to initiation of adjuvant therapy), and every three months thereafter.

SUMMARY:
The purpose of this study is to determine how circulating tumor DNA (ctDNA), a sign of minimal residual disease (MRD), is detectable after surgery in patients with early HR+/HER2- breast cancer that has spread to 1-3 lymph nodes. Researchers aim to understand if ctDNA detection can identify patients at higher risk of recurrence and guide better treatment decisions. A key aspect is the inclusion of a dedicated cohort of African American/Black women, a group underrepresented in molecular residual disease (MRD) research despite experiencing more aggressive breast cancers. This study will correlate ctDNA results with treatment patterns (radiotherapy, systemic therapy) and outcomes (recurrence-free and overall survival) in both non-African American and African American participants.

DETAILED DESCRIPTION:
Ultimately, the goal is to improve treatment strategies for this patient population. Detecting minimal residual disease (MRD) is a promising approach to identifying patients at increased risk of recurrence after definitive therapy, who may benefit from the escalation of their treatment and remain potentially curable with effective local and systemic therapy. Circulating tumor DNA (ctDNA), found in blood plasma, has recently emerged as a noninvasive approach for disease monitoring and detecting MRD through tracking tumor mutations. Nodal involvement is correlated with ctDNA positivity across multiple cancer types, and therefore, the use of ctDNA may capture patients who are more likely to have additional involvement of unresected axillary lymph nodes and can benefit from additional adjuvant therapies. One goal of this project is to investigate the clinical utility of using ctDNA as a biomarker to help tailor adjuvant radiation and systemic therapy in breast cancer (BC) patients with nodal disease, especially luminal subtype N1 BC, a group for which there is limited data available regarding the best treatment approach. As such, the primary objective of this study is to evaluate the prevalence of ctDNA-based MRD status in all patients by defining the proportion of patients with MRD-only recurrence post-operatively. Tumor tissue will be collected at surgery for genetic analysis. Blood samples for ctDNA testing will be taken at enrollment every three months. ctDNA results will be kept from treating physicians. Researchers will retrospectively analyze the relationship between ctDNA levels, administered treatments, and cancer recurrence.

A dedicated cohort of this study will enroll only African American/Black patients with early-stage, node-positive breast cancer of any subtype, who proceeded to surgery as their first treatment modality. The rationale for this cohort is to increase diversity in genomic research in Black populations, where more aggressive breast cancers are diagnosed, and non-invasive methods could provide novel insights for cancer treatment. There is a paucity of data on ctDNA prevalence and dynamics in Black patients with breast cancer, and this will be the first study of its kind to study ctDNA in Black patients. This study will provide information on ctDNA prevalence in early-stage breast cancer with 1-3 positive lymph nodes.

ELIGIBILITY:
In order to participate in this study, a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

1. Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
2. Subjects are willing and able to comply with study procedures based on the judgment of the investigator.
3. Age ≥ 18 years at time of consent.
4. Subject must have had surgical intervention and must have sufficient archival specimens from either the primary tumor or a lymph node for ctDNA assay development, as specified in the lab manual.

Exclusion Criteria:

1. Subjects must not have had prior neoadjuvant therapy.
2. Evidence of metastatic disease in imaging.
3. N1 mic or isolated tumor cells in the lymph nodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants have post-operative circulating tumor DNA (ctDNA) positive | Baseline
  Circulating tumor DNA (ctDNA) will be tested and a number of participants who were tested for positive ctDNA status. Post-operative ctDNA status will be categorized as either detectable or undetectable.

SECONDARY OUTCOMES:
Number of participants have circulating tumor DNA (ctDNA) positive in Cohort 1 | Baseline
  Circulating tumor DNA (ctDNA) will be tested and a number of participants who were tested for positive ctDNA status. ctDNA status will be categorized as either detectable or undetectable in Cohort1.

OTHER OUTCOMES:
Number of participants have circulating tumor DNA (ctDNA) positive in Cohort 2 | Baseline
  Circulating tumor DNA (ctDNA) will be tested and a number of participants who were tested for positive ctDNA status. ctDNA status will be categorized as either detectable or undetectable in Cohort2.
Number of participants have circulating tumor DNA (ctDNA) positive at 12 months | 12 months
  Circulating tumor DNA (ctDNA) will be tested at 12 month and a number of participants who were tested for positive ctDNA status. ctDNA status will be categorized as either detectable or undetectable at 12 months from the time of surgery, vs otherwise in cohorts 1 and 2.
ctDNA clearance after systemic adjuvant chemotherapy in cohorts 1 and 2 | Up to 6 months
  ctDNA clearance after systemic adjuvant chemotherapy in cohorts 1 and 2 participants with ctDNA positivity post-operatively will be defined as the proportion of participants who convert from ctDNA positive to negative after completion of adjuvant chemotherapy if indicated.
ctDNA clearance after adjuvant radiation therapy in cohorts 1 and 2 | Up to 12 months
  ctDNA clearance after adjuvant radiation therapy in cohorts 1 and 2 participants with ctDNA positivity post-operatively will be defined as the proportion of participants who convert from ctDNA positive to negative after completion of adjuvant radiation therapy, if indicated.
Recurrence-free survival | Up to 12 months
  Recurrence-free survival, defined as the time from surgery to when there is evidence of cancer recurrence, will be calculated for cohorts 1 and 2.
Overall survival | Up to 12 months
  Overall survival, defined as the time from surgery to the time of death, will be calculated for cohorts 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Yara Abdou, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials